CLINICAL TRIAL: NCT04669288
Title: AZithromycin Therapy in Preschoolers With a Severe Wheezing Episode Diagnosed at the Emergency Department (AZ-SWED)
Brief Title: AZithromycin Therapy in Preschoolers With a Severe Wheezing Episode Diagnosed at the Emergency Department
Acronym: AZ-SWED
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The AZ-SWED trial was stopped by the National Heart, Lung, and Blood Institute (NHLBI) due to futility
Sponsor: University of Arizona (Other)
Collaborators: University of Utah (Other); Emory University (Other); Morgan Stanley Children's Hospital (Other); University of Pittsburgh (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Children's Hospital of Philadelphia (Other); Children's Hospital Medical Center, Cincinnati (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Fernando Martinez, Regents' Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UG3HL147016 (NIH)
Record Dates: First submitted 2020-12-02; First posted 2020-12-16 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Asthma; Wheezing
Keywords: Wheezing Lower Respiratory Illness (WLRI)
MeSH Terms: conditions — Asthma; Respiratory Sounds | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: This Phase III trial is designed as a parallel group, placebo-controlled, double-blind, randomized, multi-center evaluation of AZ for the treatment of acute wheezing episodes. This short-term study has three planned visits. All enrolled patients will participate on the Day 0 visit for screening, the informed consent process, enrollment, randomization and dispensing. A sub-group of 370 randomly selected patients will participate in two follow-up visits on Day 5 - 8 and Day 14 - 21 where they will be tested for antibiotic resistance.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Equal allocation randomization tables will be provided by the Data Coordinating Center (DCC) to the central research pharmacy. The central research pharmacy will prepare consecutively numbered study kits according to the randomization schedule. Study kits will be sent to the clinical sites.
  Study products will be labeled with numerical codes that will maintain allocation concealment. Blinding/labeling of study medication bottles will be completed at the site pharmacy prior to dispensing to the patient.
  Randomization tables will be created at the Data Coordinating Center using permuted-block randomization stratified by clinical site and baseline severity of symptoms. Permuted blocks of random lengths 2, 4, and 6 will be used. The randomization number will be recorded in the database.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment - Active (Active Comparator): Eligible patients will be randomly assigned to one of two treatment groups (1:1) and one arm will be administered the active drug per the randomization schedule. Study medication will be provided to parents/guardians, along with instructions, for home-based administration. The first dose of the study medication will be administered before discharge from the ED.
  Interventions: Drug: Azithromycin
- Treatment - Placebo (Placebo Comparator): Eligible patients will be randomly assigned to one of two treatment groups (1:1) and one arm will be administered placebo per the randomization schedule. Study medication will be provided to parents/guardians, along with instructions, for home-based administration. The first dose of the study medication will be administered before discharge from the ED.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — oral azithromycin (12 mg/kg per day for 5 days)
  Local investigational drug pharmacies will be provided with active study medication (azithromycin) from a central pharmacy. Azithromycin will be reconstituted with water at the local pharmacy, and will resemble placebo with regards to appearance, flavor, consistency and packaging.
  Arms: Treatment - Active
Drug: Placebo — oral placebo (12 mg/kg per day for 5 days)
  Local investigational drug pharmacies will be provided with placebo from a central pharmacy. Placebo will be reconstituted with water at the local pharmacy, and will resemble azithromycin with regards to appearance, flavor, consistency and packaging.
  Arms: Treatment - Placebo

SUMMARY:
AZ-SWED is a parallel group, double blind, placebo control efficacy clinical trial with two separate hypotheses. The trial will compare the 5-day outcome of preschool children presenting to an Emergency Department (ED) with an acute, severe wheezing episode and treated with either once daily oral Azithromycin (12 mg/kg/day for 5 days) or placebo. The AZ-SWED researchers will make separate comparisons in children in whom specific pathogenic bacteria are isolated from nasopharyngeal swabs, and in those in whom they are not isolated. The primary outcome will be the Asthma Flare-up Diary for Young Children (ADYC), a validated instrument that caregivers will transmit electronically daily after discharge from the ED. Families will be contacted daily during the five-day treatment to collect the ADYC, and to assess compliance and complications. A randomly chosen subset of enrolled children will participate in two follow-up visits 5-8 days and 14-21 days after visit 1 to assess development of resistance to study drug and treatment response related changes in the airway microbiome.

DETAILED DESCRIPTION:
This Phase III trial is designed as a parallel group, placebo-controlled, double-blind, randomized, multi-center evaluation of AZ for the treatment of acute wheezing episodes. The study will recruit eligible patients from an estimated six EDs and enroll up to 2,000 patients. We will test two primary hypotheses: 1) AZ (12 mg/Kg/day) given for 5 days to preschool children with severe acute wheezing and harboring any of three specific pathogenic bacteria (H influenzae, M catarrhalis, or S pneumonia) in their nasopharynx will decrease the severity of the acute episode; and 2) AZ given on an identical schedule and dose will decrease the severity of wheezing episodes in children who do not harbor any of these three pathogenic bacteria in their nasopharynx. We will also explore whether variants in the genes encoding for Cadherin Related Family Member 3 (CDHR3), Interleukin-8 (IL-8) and in the 17q asthma-related gene cluster predict response to AZ.

This short-term study has three planned visits. All enrolled patients will participate on the Day 0 visit for screening, the informed consent process, enrollment, randomization, treatment initiation and dispensing drug. A sub-group of 370 randomly selected patients will participate in two follow-up visits on Day 5 - 8 and Day 14 - 21 where they will be tested for antibiotic resistance. The primary outcome will be the sum of the Asthma Flare-up Diary for Young Children (ADYC) score, a validated instrument completed by the parent or guardian of the enrolled children during the 5-day treatment period. Secondary outcomes will include (1) ED length of stay (2) hospital length of stay, and (3) return ED visits or hospitalizations within 72 hours after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 months to <60 months.
* The presence of expiratory wheezing as ascertained by a physician or nurse practitioner at admission to the ED.
* A Pediatric Respiratory Assessment Measurement (PRAM) score of greater than or equal to 4 at any time during the ED admission.

Exclusion Criteria:

* Presence of acute infection that requires systemic antibiotics, as determined by the physician.
* Current or previous use of systemic antibiotics within the last 2 weeks.
* Current or previous use of a steroid for wheezing within the last 2 weeks.
* Suspected foreign body induced aspiration during the last 2 weeks.
* A known systemic illness (other than allergy) including but not limited to:

  * Recurrent seizures
  * Gastroesophageal reflux (GER) requiring medical treatment
  * Major congenital anomalies
  * Physical and intellectual delay
  * Cerebral palsy
  * A history of chest surgery
  * Tuberculosis or other chronic infections
  * Primary or secondary immunodeficiency
  * Gastrointestinal malformation or disease
  * Cardiac disorder (except for a hemodynamically insignificant atrial septal defect (ASD), ventricular septal defect (VSD) or benign heart murmur)
* Born at less than 36 weeks estimated gestational age.
* Received oxygen for more than 5 days in the neonatal period, or received invasive mechanical ventilation.
* Significant developmental delay / failure to thrive, defined as a child plotting less than 3rd percentile.
* Any chronic lung disease.
* The study intervention poses undue risk to patient in the opinion of the treating physician
* Known sensitivity or allergy to AZ.
* Participation in the evaluation of a drug or medical device currently or within the last 30 days.
* Previous enrollment into this trial.
* Inability of the parent or guardian to speak English or Spanish.
* Positive PCR or antigen test for COVID-19 from hospital/doctor's office/testing center within the past 30 days.

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 840 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Asthma Flare-up Diary for Young Children | 5 day course of azithromycin
  The Asthma Flare-up Diary for Young Children (ADYC) is a validated instrument that consists of a 17-item questionnaire scored from 1 (best) to 7 (worst). The parent or guardian of the enrolled child (up to 60 months of age) will fill out the diary daily for 5 days, starting from the first day following the first dose of Azithromycin (AZ). The cumulative score at the end of 5 days will be used to assess response to the intervention (e.g. time to exacerbation, acute-care visit, hospitalization and no wheeze), with a higher score indicating a worse outcome.

SECONDARY OUTCOMES:
Length of Stay | 72 hours after randomization
  Secondary outcomes will include (1) ED length of stay (2) hospital length of stay, and (3) return ED visits or hospitalizations.
Number of participants that develop Azithromycin resistant organisms | 21 days after randomization
  Presence of azithromycin-resistant organisms will be assessed at baseline, and again at two follow-up visits 5-8 days and 14-21 days after enrollment in a randomly selected subset of trial subjects. A total of 370 subjects will be selected for this follow-up. Subjects in whom resistance is detected at baseline will not be included in the analysis of development of bacterial resistance at follow-up. Among subjects that are negative for bacterial resistance at baseline, follow-up resistance will be tabulated by treatment. The absolute risk diﬀerence, together with a 95% one-sided conﬁdence interval, will be used to summarize treatment diﬀerence. Participants who harbor or do not harbor the three pathogenic bacteria will be included in these analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Martinez, MD, Principal Investigator — University of Arizona; Kurt Denninghoff, MD, Principal Investigator — University of Arizona; Charlie Casper, PhD, Principal Investigator — University of Utah
Locations (8):
- United States (8):
  - Children's Healthcare of Atlanta, Emory University, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of New York Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
After subject enrollment and follow up have been completed, the DCC may prepare a final study database for analysis. A releasable database will be produced and completely de-identified in accordance with the definition provided in the Health insurance Portability and Accountability Act (HIPAA). HIPAA will be recoded in a manner that will make it impossible to deduce or impute the specific identity of any patient. The database will not contain any institutional identifiers. This releasable database will be forwarded to the Biologic Specimen and Data Repository Information Coordinating Center (BIOLINCC) or, in case AZ-SWED samples and data are not deposited in BIOLINCC, to users in electronic form, in accordance with policies determined by the investigators and funding sponsors.